CLINICAL TRIAL: NCT03408223
Title: Total Marrow and Lymphoid Irradiation and Chemotherapy Prior to Allogeneic Hematopoietic Cell Transplant for High-Risk Acute Leukemia
Brief Title: Total Marrow and Lymphoid Irradiation and Chemotherapy for High-Risk Acute Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Chen Hu, Principal Investigator, Affiliated Hospital to Academy of Military Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LouX02
Record Dates: First submitted 2017-12-24; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Whole-Body Irradiation; Lymphatic Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total body irradiation (Active Comparator): Patient receives preparative therapy including cyclophosphamide and total body irradiation (TBI) of 10 Gy on Days -4 through -1, and starts immunosuppressive therapy using cyclosporine or tacrolimus, methotrexate-based prophylaxes, followed by peripheral blood stem cell transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Radiation: total body irradiation
- total marrow and lymphoid irradiation (Experimental): Patient receives preparative therapy including cyclophosphamide and total marrow and lymphoid irradiation of 12-20 Gy on Days -8 through -2, and starts immunosuppressive therapy using cyclosporine or tacrolimus, methotrexate-based prophylaxes, followed by peripheral blood stem cell transplantation and granulocyte colony-stimulating factor administration.
  Interventions: Radiation: total marrow and lymphoid irradiation

INTERVENTIONS:
Radiation: total body irradiation — Drug: Cyclophosphamide 60 mg/kg/day intravenous x 2 days pre-transplant, total dose 120 mg/kg
  Drug: Cyclosporine or tacrolimus Beginning on Day -1 pre-transplant maintaining a level of 150-250 ng/ml or 5-10 ng/ml respectively. Cyclosporine or tacrolimus dosing will be monitored and altered as clinically appropriate by physician, and discontinue at approximately day + 180 post-transplant.
  Drug: Methotrexate 15 mg/m2 intravenous on days 1, 10 mg/m2 intravenous on days 3, 6 and 11 after transplantation.
  Intervention: Total Body Irradiation Dose of 10 Gy TBI (fraction size of 5 Gy given once a day on days -2 and -1).
  Procedure: Peripheral blood stem cell transplantation product will be infused via intravenous drip on Day 0.
  Other Names: TBI
  Arms: total body irradiation
Radiation: total marrow and lymphoid irradiation — Drug: Cyclophosphamide 60 mg/kg/day intravenous x 2 days pre-transplant, total dose 120 mg/kg
  Drug: Cyclosporine or tacrolimus Beginning on Day -1 pre-transplant maintaining a level of 150-250 ng/ml or 5-10 ng/ml respectively. Cyclosporine or tacrolimus dosing will be monitored and altered as clinically appropriate by physician, and discontinue at approximately day + 180 post-transplant.
  Drug: Methotrexate 15 mg/m2 intravenous on days 1, 10 mg/m2 intravenous on days 3, 6 and 11 after transplantation.
  Intervention: Total Marrow and Lymphoid Irradiation Dose of 12-20 Gy TMLI (fraction size of 4 Gy given once a day).
  Procedure: Peripheral blood stem cell transplantation product will be infused via intravenous drip on Day 0.
  Other Names: TMLI
  Arms: total marrow and lymphoid irradiation

SUMMARY:
RATIONALE: Giving chemotherapy and total marrow and lymphoid irradiation before allogeneic hematopoietic cell transplant helps stop the growth of leukemia cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may achieve brand new hematopoietic recovery. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells, resulting in graft versus-host disease.

PURPOSE: This study is to evaluate the toxicity and efficacy of total marrow and lymphoid irradiation conditioning when given together with combination chemotherapy and allogeneic peripheral blood stem cell transplant in treating patients with high-risk acute leukemia.

DETAILED DESCRIPTION:
Patient receives preparative therapy including cyclophosphamide and total body irradiation (TBI) of 10 Gy or total marrow and lymphoid irradiation (TMLI) of 12-20 Gy, and starts immunosuppressive therapy using cyclosporine or tacrolimus, methotrexate-based prophylaxes, followed by peripheral blood stem cell transplantation and granulocyte colony-stimulating factor administration.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk acute myelogenous leukemia or acute lymphocytic leukemia based on clinical and biological characteristics, which including but not limited to poor response to induction therapy and relapse or beyond second remission.
2. Karnofsky performance status (KPS) >= 70%
3. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
4. All candidates for this study must have a prepared allogeneic stem cell donor, including human leukocyte antigen matched or partially mismatched donor
5. A cardiac evaluation with an electrocardiogram showing no ischemic changes or abnormal rhythm and an ejection fraction of >= 50% established by multi gated acquisition scan (MUGA) or echocardiogram
6. Patients must have a serum creatinine of less than or equal to 1.3 mg/dL or creatinine clearance >70 ml/min
7. Hepatic: bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Alkaline phosphatase (ALP) < 5 x upper limit of normal (ULN)
8. Pulmonary function: Carbon Monoxide Diffusing Capacity corrected (DLCOcorr) > 50% of normal, (oxygen saturation [>92%] can be used in child where pulmonary function tests (PFT's) cannot be obtained)
9. The time from the end last induction or re-induction attempt should be greater than or equal to 14 days
10. All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Active uncontrolled infection at time of enrollment or documented fungal infection within 3 months
2. Evidence of Human immunodeficiency virus (HIV) infection
3. Prior myeloablative transplant within the last 6 months
4. Prior radiation therapy that would exclude the use of TMLI
5. Relapsed patients who have undergone autologous or allogeneic hematopoietic stem cell transplantation previously

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity, scored on National Cancer Institute Common Terminology Criteria version 4.03 | Up to 100 days after stem cell infusion
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen.
Progression-Free Survival (PFS) | The time from start of protocol therapy to death, relapse/progression, or last follow-up, whichever comes first, assessed up to 2 years
  Calculated using the Kaplan-Meier method. The cumulative incidence of relapse/progression will be calculated as a competing risk using the Gray method.

SECONDARY OUTCOMES:
Incidence of transplantation-related mortality | 6 months
  In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Incidence of grade II-IV acute graft-versus-host disease (GVHD) after transplantation | Day +100
  Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Incidence of chronic GVHD after transplantation | 1 Year
  Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host.
Incidence of relapse after transplantation | 1 year and 2 years
  The return of disease after its apparent recovery/cessation.
Menstrual recovery after transplantation | 1 year and 2 years
  The percentage of female patients who have resumed menses is usually considered as related to ovarian function.
Overall survival after transplantation | The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer.
  1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hu Chen, M.D., Ph.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences (307 Hospital of PLA)
Locations (1):
- Affiliated Hospital to Academy of Military Medical Sciences (307 Hospital of PLA), Beijing, Beijing Municipality, China